CLINICAL TRIAL: NCT03335397
Title: Interactive Learning Strategies Using M-learning for Improving Professional Competencies in Health Sciences
Brief Title: M-learning to Improve Professional Competencies in Health Sciences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Irene Cantarero Villanueva, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID 16-54
Record Dates: First submitted 2017-10-31; First posted 2017-11-07 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Education
Keywords: education; health science; app; m-learning
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-learning group (Experimental): Participants receive mobile app (m-learning application) with interactive content (quiz).
  Interventions: Device: M-learning application
- Control group (Other): Participants receive traditional learning process (books, journals available in the University library).
  Interventions: Other: Traditional learning process

INTERVENTIONS:
Device: M-learning application — Mobile application with interactive contents available for android platform and Apple's operating system.
  Arms: M-learning group
Other: Traditional learning process — Traditional content available in university library.
  Arms: Control group

SUMMARY:
The aim of this study is to investigate whether a mobile application is useful for improving knowledge about professional competencies in students enrolled in Health Sciences degrees.

DETAILED DESCRIPTION:
The learning environment in Higher Education as well as autonomous work of students, mobile technology is increasingly present due to the mass use of mobile devices and the development of high speed in data transmission, which provides today the possibility of being able to access in real time a great amount of information.

M-learning is defined as the ability to access educational resources, tools and materials using a mobile device anytime and anywhere.

Considering the advantages of this technology, m-learning can be a real option to the traditional teaching-learning method by encouraging the active participation of students in their own learning process.

Therefore, this educational innovation study aims to evaluate the effectiveness and the use of a mobile application as a complementary learning strategy in interactive format for the acquisition of professional competencies in Health Sciences.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Access last generation mobile phone
* Enroll 1º course Health Sciences degrees
* Basic english knowledge

Exclusion Criteria:

* Prior experience in Fundaments subject (second enrolment or more not allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Multiple-choice questions | Change scores: Baseline, 2-week intervention
  The knowledge gain is evaluated using a 20-item multiple-choice questions (MCQs), a learning assessment tool with a minimum of 0 points and maximum of 10 points, with higher values represent a better outcome.

SECONDARY OUTCOMES:
Instructional Materials Motivation Survey | 2-week intervention
  The level of learning motivation is evaluated using Instructional Materials Motivation Survey (IMMS). The IMMS consists of four domains: attention, relevance, confidence, and satisfaction, with a total of 36 questions on a 5-point Likert scale. Possible scores range from 36 to 180, with a higher score indicative of a higher level of learning motivation.
Satisfaction survey questionnaire | 2-week intervention
  Satisfaction is measured using Likert scale scores for different items, with higher values represent a better outcome.
Profile of Mood States | Change scores: Baseline, 2-week intervention
  The Profile of Mood States (POMS) questionnaire is a measure of emotional state. It contains 65 items assessing mood state, which are grouped into six subscales: tension-anxiety, depression-dejection, anger-hostility, vigour-activity, fatigue-inertia and confusion-bewilderment. The score rate is a Likert scale (not at all: 0; a little: 1; moderately: 2; quite a lot: 3; extremely: 4).

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cantarero-Villanueva, PhD, Principal Investigator — Health Science Faculty. University of Granada, Granada (Spain)
Locations (1):
- University of Granada, Granada, Spain

REFERENCES:
- [Derived] Lozano-Lozano M, Fernandez-Lao C, Cantarero-Villanueva I, Noguerol I, Alvarez-Salvago F, Cruz-Fernandez M, Arroyo-Morales M, Galiano-Castillo N. A Blended Learning System to Improve Motivation, Mood State, and Satisfaction in Undergraduate Students: Randomized Controlled Trial. J Med Internet Res. 2020 May 22;22(5):e17101. doi: 10.2196/17101. PMID 32441655